CLINICAL TRIAL: NCT03862040
Title: An Open-label, Multicenter, Single-arm, Phase 1 Study to Assess the Intrapulmonary Concentrations of Cefiderocol at Steady State in Hospitalized Subjects With Known or Suspected Bacterial Pneumonia on Treatment With Standard of Care Antibiotics and Requiring Mechanical Ventilation
Brief Title: Cefiderocol Concentrations in the Lungs of Hospitalized Patients With Bacterial Pneumonia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1713R2117
Expanded Access: NCT03780140 (Approved for marketing)
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Bacterial Pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — Cefiderocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cefiderocol (Experimental): All participants were receiving standard of care (SOC) antibiotic treatment for pneumonia. Forty hours after the start of SOC treatment, participants will be administered 2 g doses of cefiderocol (or renally adjusted doses) infused intravenously over 3 hours, every 8 hours (or every 6 hours for participants with augmented renal function), for an expected minimum of 3 doses and up to a total of 6 doses in participants with normal renal function and participants with mild or moderate renal impairment, and for an expected minimum of 6 doses and up to a total of 9 doses in participants with severe renal impairment.
  Interventions: Drug: Cefiderocol; Drug: Standard of Care Antibiotic

INTERVENTIONS:
Drug: Cefiderocol — Administered intravenously, at a dosage determined based on renal function.
  Other Names: S-649266)
Drug: Standard of Care Antibiotic — Standard of care antibiotic treatment for pneumonia

SUMMARY:
The primary purpose of the study is to determine the degree of penetration of cefiderocol into infected lung tissue in hospitalized adults with bacterial pneumonia who are being mechanically ventilated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older at the time written informed consent is obtained
2. Subject has provided written informed consent or informed consent has been provided by subject's legally authorized representative
3. Subject has a diagnosis or suspicion of bacterial pneumonia (even if later known that the subject does not have bacterial pneumonia, discontinuation of the study is not necessary)
4. Subject is hospitalized and receiving standard of care antibiotic treatment for pneumonia
5. Subject is mechanically ventilated or expected to be mechanically ventilated at least 48 hours (or 72 hours for subjects with severe renal impairment) after the first dose of cefiderocol
6. Subject has a life expectancy of at least 3 weeks from the Screening visit
7. Subject is male (no contraception required) or female and meets 1 of the following criteria:

   1. Surgically sterile (has had a hysterectomy and/or bilateral oophorectomy, or a bilateral salpingectomy or tubal ligation for the purpose of contraception for at least 6 weeks with appropriate documentation of such surgery)
   2. Postmenopausal (defined as older than 45 years of age with cessation of regular menstrual periods for at least 6 months and a follicle-stimulating hormone level of > 40 mIU/mL, or amenorrhea for at least 12 months)
   3. Of childbearing potential and using combined (estrogen and progestogen) or progestogen-only hormonal contraception associated with inhibition of ovulation (including oral, intravaginal, injectable, implantable, and transdermal contraceptives), or an intrauterine device (IUD), or intrauterine hormone-releasing system for the entire duration of the study
   4. Of childbearing potential and practicing abstinence as a preferred and usual life style and/or agrees to continue practicing abstinence from Screening for the entire duration of the study
   5. Of childbearing potential and whose sole heterosexual partner has been successfully vasectomized and agrees to not have other heterosexual partners for the entire duration of the study

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Subject has a chemical pneumonia that does not require antibiotic treatment (including aspiration of gastric acid, inhalation injury). The term chemical pneumonia refers to the aspiration of substances that are toxic to the lower airways causing chemical burn and injuries in the airway.
2. Subject has a history of any moderate or severe hypersensitivity or allergic reaction to any β-lactam (Note: for β-lactams, a history of a mild rash followed by uneventful re-exposure is not a contraindication to enrollment)
3. Subject has extensive cystic lesion(s) or severe structural abnormality (eg, cystic fibrosis, emphysema, cystic lesions of sarcoidosis or tuberculosis, postobstructive pneumonia due to lung cancer, etc) of the lung that hinders recovery of bronchoalveolar lavage fluid (BALF)
4. Subject is receiving peritoneal dialysis
5. Subject has severe renal impairment requiring hemodialysis (HD) or end-stage renal disease requiring HD
6. Subject is in refractory septic shock defined as persistent hypotension despite adequate fluid resuscitation or despite vasopressive therapy at Screening
7. Subject is a female who has a positive pregnancy test at Screening or who is lactating
8. Subject has received another investigational drug within 30 days prior to Screening
9. Subject has previously participated in this clinical study and has received at least 1 dose of cefiderocol within 7 days
10. Subject has any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (7):
- United States (7):
  - Anschutz Medical Campus, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida, Jacksonville, Florida
  - U Miami Health Tower, Miami, Florida
  - North Western University, Chicago, Illinois
  - Creighton University, Omaha, Nebraska
  - Weill Cornell Medical College, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 3 sites in the United States. Seven adults with known or suspected bacterial pneumonia being treated with standard of care (SOC) antibiotics and requiring mechanical ventilation were enrolled.
Groups:
- Cefiderocol: Participants received 2 g cefiderocol (or renally adjusted doses) every 8 hours (or every 6 hours for participants with augmented renal function), administered by intravenous infusion over 3 hours for a total of 3 to 6 doses.
Period: Overall Study
Arm/Group | Cefiderocol
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cefiderocol
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5
  Black or African American | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Cefiderocol in Epithelial Lining Fluid
Description: Samples for determination of cefiderocol concentrations in the epithelial lining fluid (ELF) were collected by bronchoalveolar lavage (BAL) procedure on the inflamed section of the lung (ie, a lobe where pneumonia was expected to be present based on chest radiologic imaging) after multiple doses of cefiderocol sufficient to approximate steady state concentrations in blood. The ELF sample for the determination of cefiderocol concentrations was collected at 3 hours after the start of administration of cefiderocol for the first 4 enrolled participants and at 2 hours after the end of infusion for the following 3 participants.
  Cefiderocol concentrations were determined using liquid chromatography/tandem mass spectrometry (LC/MS/MS), with a lower limit of quantification of cefiderocol in ELF of 0.005 μg/mL. Cefiderocol concentrations in ELF were calculated using cefiderocol concentrations in BAL, adjusted by the ratio of urea concentrations in blood and BAL.
Time Frame: At the third dosing (or sixth dosing for participants with severe renal impairment; 16 or 40 hours after first dose, respectively), at 3 hours after the start of the infusion or 2 hours after the end of infusion.
Population: All participants who received at least 1 dose of cefiderocol and who had at least 1 evaluable concentration of cefiderocol in bronchoalveolar lavage fluid.
Measure: Geometric Mean (Full Range); unit: μg/mL
Arm/Group | Cefiderocol
Number analyzed (Participants) | 7
μg/mL
  3 hours after start of infusion: number analyzed (Participants) | 4
  3 hours after start of infusion | 7.63 [3.10 to 20.7]
  2 hours after end of infusion: number analyzed (Participants) | 3
  2 hours after end of infusion | 10.4 [7.19 to 15.9]

2. Primary Outcome: Ratio of the Concentration of Cefiderocol in Epithelial Lining Fluid Relative to Plasma
Description: The concentration of cefiderocol in ELF to plasma ratio (RC,E/P) represents the penetration of cefiderocol into infected lung tissue.
  ELF and plasma cefiderocol concentrations were determined using liquid chromatography/tandem mass spectrometry (LC/MS/MS). The lower limit of quantification of cefiderocol in plasma and ELF was 0.1 μg/mL and 0.005 μg/mL, respectively.
Time Frame: At the third dosing (or sixth dosing for participants with severe renal impairment; 16 or 40 hours after start of the first dose, respectively), at 3 hours after the start of the infusion or 2 hours after the end of infusion.
Population: All participants who received at least 1 dose of cefiderocol and who had at least 1 evaluable concentration of cefiderocol in bronchoalveolar lavage fluid. Cefiderocol concentration was measured 3 hours after the start of the infusion in the first 4 enrolled participants and 2 hours after the end of infusion in the following 3 participants.
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | Cefiderocol
Number analyzed (Participants) | 7
ratio
  3 hours after start of infusion: number analyzed (Participants) | 4
  3 hours after start of infusion | 0.0893 [0.0379 to 0.178]
  2 hours after end of infusion: number analyzed (Participants) | 3
  2 hours after end of infusion | 0.231 [0.187 to 0.347]

ADVERSE EVENTS:
Time Frame: From the start of the first infusion of cefiderocol up to 7 days after last dose, up to 9 days.
Arm/Group | Cefiderocol
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cefiderocol (N=7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hyperchloraemia (Metabolism and nutrition disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Bacteriuria (Infections and infestations) | 1
Blood urea increased (Investigations) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Wound dehiscence/ (Injury, poisoning and procedural complications) | 1
Implant site dehiscence (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT03862040/SAP_000.pdf
  • Study Protocol (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03862040/Prot_001.pdf